CLINICAL TRIAL: NCT00198146
Title: PD Initiated/Prevention of Diabetes Progression Trial (PDPT) ZEN119
Brief Title: Prevention of Diabetes Progression Trial (PDPT)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indiana University School of Medicine (Other)
Collaborators: Pescovitz, Mark D., M.D. (Individual); Roche Pharma AG (Industry); Facet Biotech (Industry)
Organization: Indiana University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9910-34
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2020-08-11 (Actual); Status verified 2005-09

CONDITIONS: Newly Diagnosed With Type 1 Diabetes
MeSH Terms: interventions — Daclizumab

INTERVENTIONS:
Drug: Zenapax

SUMMARY:
The primary purpose of this study is to determine the efficacy and safety of daclizumab in preventing the progression of diabetes in children who have just been diagnosed with type I diabetes. Additional purposes of the study are to investigate the amount of drug in the children, how quickly it is eliminated from the blood, and analyze the effect of the drug on the immune reaction to diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed type 1 diabetes without previous insulin or oral hypoglycemic therapy.
* ages 2 to 40 years at diagnosis
* enroll within 3 months of diagnosis
* test positive for at least one of the biochemical autoantibodies (ICA-512, GAD 65 or IAA) prior to enrolling

Exclusion Criteria:

* Previous treatment with an anti-IL-2 directed monoclonal antibody or any other investigational agent that would interfere with the ability to evaluate the safety and efficacy of daclizumab.
* Other immunosuppressive drugs including, but not limited to, corticosteroids, cyclosporine, tacrolimus, rapamycin, mycophenolate mofetil, or azathioprine.
* Active significant infection
* Limited life expectancy because of disease other than diabetes
* Pregnancy

Ages: 2 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40
Dates: Start 2000-07; Primary Completion 2007-02-23 (Actual); Study Completion 2007-02-23 (Actual)

PRIMARY OUTCOMES:
Area under the curve, Glucagon Stimulation Testing for c-peptide measurements at 0, +6min and +10min intervals over 2 years

SECONDARY OUTCOMES:
HbA1c
Insulin requirements (units/kg/day)

CONTACTS AND LOCATIONS:
Overall Officials: Mark D Pescovitz, M.D., Principal Investigator — Indiana University - Riley Hospital for Children
Locations (1):
- Indiana University - Riley Hospital for Children, Indianapolis, Indiana, United States